CLINICAL TRIAL: NCT00914368
Title: TOPAS-1, A Pharmacodynamic Phase II Study of Clopidogrel P2Y12 Platelet Inhibition
Brief Title: Tailoring Of Platelet Inhibition to Avoid Stent Thrombosis
Acronym: TOPAS-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Lars Wallentin, MD, PhD. Professor Cardiology, UCR, Uppsala University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: U-08-002
Record Dates: First submitted 2009-05-29; First posted 2009-06-05 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2009-09

CONDITIONS: Coronary Artery Disease; Myocardial Infarction; Stent Thrombosis; Heart Diseases; Acute Coronary Syndrome
Keywords: Platelet Aggregation Inhibitors; Aspirin; Clopidogrel; Pathologic Processes; Disease; Therapeutic Uses; Syndrome; Hematologic Agents; Cardiovascular Diseases; Pharmacologic Actions
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Heart Diseases; Acute Coronary Syndrome; Pathologic Processes; Disease; Syndrome; Cardiovascular Diseases | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Patients with previously experienced stent thrombosis while on dual antiplatelet treatment within 6 months after coronary stenting for coronary artery disease
  Interventions: Drug: Clopidogrel
- 2 (Active Comparator): Patients with previously experienced myocardial infarction while on dual antiplatelet treatment within 6 months after coronary stenting for coronary artery disease
  Interventions: Drug: Clopidogrel
- 3 (Active Comparator): Patients without previously experienced myocardial infarction or stent thrombosis 6 within months after coronary stenting for coronary artery disease(matched controls for group 1 and 2)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Patients not already on clopidogrel treatment a loading dose of clopidogrel 600 mg followed by a maintenance dose of 75 mg once daily will be administered.
  Other Names: Plavix

SUMMARY:
The primary objective of this study is to establish a cut off level of platelet inhibition that separates patients with or without previous stent occlusion with acute clinical onset while on aspirin and clopidogrel treatment within 6 months after coronary stenting for coronary artery disease.

DETAILED DESCRIPTION:
To establish cut off levels of platelet inhibition using ADP-induced P2Y12-receptor mediated platelet aggregation using Accumetrics VerifyNow P2Y12 assay (PRU) and Vasodilator-stimulated phosphoprotein (VASP, PRI %)for patients with experienced stent occlusion with acute clinical onset and/or myocardial infarction within 6 months after coronary stenting for coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written informed consent.
* Male or female patients above 18 years old.
* Previous PCI and coronary stenting for coronary artery disease
* Previous (after coronary stenting) or current dual antiplatelet treatment (aspirin 75 mg once daily (o.d) and clopidogrel 75 mg o.d). All patients need to be on treatment with aspirin 75 mg once daily at least seven days prior to enrollment.
* Experienced one of the following alternatives:

  * Stent thrombosis within 6 months of PCI while on dual antiplatelet treatment; OR
  * Experienced MI within 6 month after coronary stenting while on dual antiplatelet treatment; OR
  * No experience of stent thrombosis or MI for at least 6 months and until visit 1 (matched control)

Exclusion Criteria:

General exclusion criteria:

1. Women who are known to be pregnant, who have given birth within the past 90 days, or who are breastfeeding.
2. Any condition or laboratory findings which in the opinion of the Investigator makes the patient unsuitable for inclusion
3. Enrolled in either another investigational drug study or in another investigational study of an approved drug within 30 days prior to Visit 1 of the current study.
4. Known allergies or intolerance to aspirin and/or thienopyridines (clopidogrel or ticlopidine).
5. Significant active neuropsychiatric disease, alcohol abuse or drug abuse, in the investigator's opinion.
6. UCR or Accumetrics employees or investigator site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.

   Cardiovascular Exclusion Criteria:
7. Subjects with unstable coronary artery disease, defined as new, increased, or rest angina at screening.
8. Subjects with significant hypertension (systolic blood pressure > 180 mm Hg or diastolic blood pressure >110 mmHg) at the time of screening.

   Bleeding Risk Exclusion Criteria:
9. Any known contraindication to treatment with an anticoagulant or antiplatelet agent.
10. Prior history or presence of significant bleeding disorders (for example,hematemesis, melena, severe or recurrent epistaxis, hemoptysis, hematuria, or intraocular bleeding)
11. Prior history or clinical suspicion of cerebral vascular malformations
12. Prior history of abnormal bleeding tendency (i.e. prolonged bleeding on dental extraction, tonsillectomy, or previous surgical procedure).
13. Personal or family history of coagulation or bleeding disorders.
14. Thrombocytopenia (platelet count < 100,000/mm3) or thrombocytosis (platelet count > 500,000/mm3).
15. History of major surgery, severe trauma, organ biopsy within 3 months prior to enrollment.
16. Any planned surgical procedure within 20 days following inclusion.
17. The use (or planned use) of other antiplatelet agents (besides aspirin and clopidogrel), anticoagulant or fibrinolytic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
VerifyNow P2Y12 (PRU) | Within 6 months

SECONDARY OUTCOMES:
VASP (PRI, %) | Within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wallentin, MD, PhD, Principal Investigator — Uppsala University, Uppsala Clinical Research Center
Locations (1):
- Uppsala Clinical Research Center, Uppsala, Sweden